CLINICAL TRIAL: NCT05074563
Title: Enhancing Resilience in the Nursing Workforce in the COVID-19 Environment: Transitioning From Face-to-face to Online Learning
Brief Title: Resilience Enhancement Online Training for Nurses (REsOluTioN) Trial
Acronym: REsOluTioN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford Brookes University (Other)
Responsible Party: Principal Investigator, Dr Cathy Henshall, Reader, Faculty of Health and Life Sciences, Oxford Brookes University, Oxford Brookes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 21/HRA/1418
Record Dates: First submitted 2021-09-23; First posted 2021-10-12 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Resilience
Keywords: Nurses; Online training; Resilience; Mentorship; Mental wellbeing
MeSH Terms: interventions — Pharmaceutical Solutions; Nurses

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Participants will not be blinded to group allocation and will complete self-reported surveys online. One of the study investigators not involved in the delivery of training or randomisation process and who will analyse the survey responses will be blinded to treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online REsOluTioN training (Active Comparator): The active comparator arm will receive access to online REsOluTioN training to enhance resilience.
  Interventions: Other: REsOluTioN (Resilience Enhancement Online Training for Nurses)
- Control (Other): The control arm will have no access to the online training.
  Interventions: Other: Control

INTERVENTIONS:
Other: REsOluTioN (Resilience Enhancement Online Training for Nurses) — The online REsOluTioN training involves virtual or face-to-face mentorship sessions and facilitated online interactive group sessions on four topics (Building hardiness and maintaining a positive outlook, Intellectual flexibility and Emotional Intelligence; Achieving life balance and enabling spirituality and Reflective and critical thinking). The training will be of four-week duration. Over the four-week period, the training will comprise 4x120 minute facilitated online group sessions; 4x30 minute independent learning activities; and eight 3:1 online mentoring sessions delivered between 30 and 60 minutes at flexible timings.
  Arms: Online REsOluTioN training
Other: Control — Nurses randomised to the control group will only be invited to take part in the pre- and post- intervention surveys, but will not use the online training. However, after completing the survey, nurses will be given the opportunity to complete the pre-work and access the facilitated sessions of the training so that they can receive their CPD certificate.
  Arms: Control

SUMMARY:
The purpose of the study is to pilot a new training which aims to foster resilience to some of the clinical and workload pressures that nurses encounter on a daily basis.

DETAILED DESCRIPTION:
Background:

Many nurses are exposed to challenges in their clinical setting on a daily basis, which often results in them experiencing stress, burnout and decreased satisfaction with their work; this can have a long term impact on the recruitment and retention rate of these nurses. This stress has intensified over the last year due to the COVID-19 pandemic. The online training being piloted in this trial has been adapted from a recent face-to-face resilience enhancement programme developed for nurses in the UK. By creating an online training, it is hoped that this intervention will be accessible to more nurses, particularly in the context of the COVID-19 pandemic.

Objectives:

The purpose of this trial is to understand whether the online training can improve levels of resilience, psychological, and wellbeing, and whether or not it has changed the way nurses experience in their work environment.

Methods:

All registered nurses working at Oxford Health NHS Foundation Trust during the COVID-19 pandemic will be invited. We intend to recruit 100 nurses who are currently working at Oxford Health NHS Foundation Trust to participate in the pilot study. Recruited nurses will be randomised to the intervention group or the control group. Nurses who are randomised to the intervention group will be invited to do the online training over a four week period. There will be the opportunity to participate in four 2 hour online facilitated sessions during the four-week training period. Nurses will also be asked to complete 30 minutes of independent pre-work ahead of each of the facilitated sessions. The sessions will cover a range of topics and will tackle areas such as building hardiness and maintaining a positive outlook; emotional intelligence and intellectual flexibility; reflective and critical thinking; enabling spirituality and achieving work-life balance. The training also involves twice weekly mentorship sessions ranging between 30 and 60 minutes.

Nurses will be invited to complete two surveys (pre- and post- intervention) which will be used to evaluate the trial outcomes and feedback on training. On completion of the post-intervention survey, nurses will receive a certificate for 10 hours of CPD. Nurses randomised to the control group will only be invited to take part in the pre- and post- intervention surveys, but will not use the online training. However, after completing the survey, nurses will be given the opportunity to complete the pre-work and access the online facilitated sessions so they can receive their CPD certificate.

Implications:

Once the training has been piloted, the effectiveness of the online training will be evaluated at national level.

ELIGIBILITY:
Inclusion Criteria:

* Any registered, non-agency nurses working at Oxford Health NHS Foundation Trust
* Willing to participate and provide signed consent

Exclusion Criteria:

* Not willing to participate and provide signed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
Resilience | Four weeks
  Brief Resilience Scale - Scores range from 1 (low resilience) to 5 (high resilience).

SECONDARY OUTCOMES:
Mental wellbeing | Four weeks
  Warwick-Edinburgh Mental Wellbeing Scale -The total score of the 14-item Warwick-Edinburgh Mental Wellbeing Scale ranges from 14-70. Higher scores indicate higher level of mental well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Cathy Henshall, PhD, Principal Investigator — Oxford Brookes University
Locations (1):
- Faculty of Health and Life Sciences, Oxford Brookes University, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Henshall C, Davey Z, Jackson D. The implementation and evaluation of a resilience enhancement programme for nurses working in the forensic setting. Int J Ment Health Nurs. 2020 Jun;29(3):508-520. doi: 10.1111/inm.12689. Epub 2020 Jan 12. PMID 31930654
- [Background] Davey Z, Jackson D, Henshall C. The value of nurse mentoring relationships: Lessons learnt from a work-based resilience enhancement programme for nurses working in the forensic setting. Int J Ment Health Nurs. 2020 Oct;29(5):992-1001. doi: 10.1111/inm.12739. Epub 2020 Jun 13. PMID 32536021
- [Background] Henshall C, Davey Z, Jackson D. Nursing resilience interventions-A way forward in challenging healthcare territories. J Clin Nurs. 2020 Oct;29(19-20):3597-3599. doi: 10.1111/jocn.15276. Epub 2020 Apr 15. No abstract available. PMID 32237252
- [Derived] Henshall C, Davey Z, Srikesavan C, Hart L, Butcher D, Cipriani A. Implementation of a Web-Based Resilience Enhancement Training for Nurses: Pilot Randomized Controlled Trial. J Med Internet Res. 2023 Feb 14;25:e43771. doi: 10.2196/43771. PMID 36787181
- [Derived] Srikesavan C, Davey Z, Cipriani A, Henshall C. Resilience Enhancement Online Training for Nurses (REsOluTioN): Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2022 Aug 3;11(8):e37015. doi: 10.2196/37015. PMID 35862692
- See also: The implementation and evaluation of a resilience enhancement programme for nurses working in the forensic setting. — https://pubmed.ncbi.nlm.nih.gov/31930654/
- See also: The value of nurse mentoring relationships: Lessons learnt from a work-based resilience enhancement programme for nurses working in the forensic setting. — https://pubmed.ncbi.nlm.nih.gov/32536021/
- See also: Nursing resilience interventions-A way forward in challenging healthcare territories. — https://pubmed.ncbi.nlm.nih.gov/32237252/